CLINICAL TRIAL: NCT07108270
Title: A Phase 2, Multicenter, Open-label, Single Arm Study of Dostarlimab Plus Carboplatin-paclitaxel Followed by Dostarlimab Monotherapy in Participants With dMMR/MSI-H Primary Advanced or Recurrent Endometrial Cancer in China (China RUBY)
Brief Title: A Study of Dostarlimab in Combination With Carboplatin-paclitaxel in Chinese Participants With Primary Advanced or Recurrent Endometrial Cancer (EC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 222258
Record Dates: First submitted 2025-08-05; First posted 2025-08-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Neoplasms, Endometrial
Keywords: Endometrial cancer; Dostarlimab; Carboplatin; Paclitaxel
MeSH Terms: conditions — Endometrial Neoplasms | interventions — dostarlimab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dostarlimab-Carboplatin-Paclitaxel followed by Dostarlimab Monotherapy (Experimental)
  Interventions: Biological: Dostarlimab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: Dostarlimab — Dostarlimab will be administered.
Drug: Carboplatin — Carboplatin will be administered.
Drug: Paclitaxel — Paclitaxel will be administered.

SUMMARY:
The goal of this clinical trial is to see how well dostarlimab works when administered with the chemotherapy drugs carboplatin and paclitaxelin in treating EC in Chinese participants. The study aims to understand the treatments effectiveness, safety, how the drugs behave in the body, and whether it causes any immune reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has histologically or cytologically proven EC with recurrent or advanced disease.
2. Participant has molecular subtype of defective mismatch repair (dMMR) or microsatellite instability high (MSI-H) determined by the central reference laboratory before study intervention.
3. Participant must have primary Stage III or Stage IV disease or first recurrent EC with a low potential for cure by radiation therapy or surgery alone or in combination, and presence of at least one target lesion per RECIST 1.1 based on Investigator's assessment and meet at least 1 of the following criteria:

   1. Has primary Stage III to IV disease and is naive to systemic anticancer therapy for EC;
   2. Has first recurrent disease and is naïve to systemic anticancer therapy for EC;
   3. Had received prior neo-adjuvant/adjuvant anticancer therapy and had a recurrence or PD ≥6 months after completing treatment (first recurrence only).
4. Participant has adequate archive tumor tissue sample for MMR/MSI status testing. If no archival tissue is available, tissue sample must be obtained before study intervention.
5. Participant is not pregnant or breastfeeding and agrees to use a highly effective contraceptive method during the study period if a woman of childbearing potential (WOCBP).
6. Participant has an Eastern Cooperative Oncology Group Performance status (ECOG PS) of 0 or 1.
7. Participant has adequate organ function, as assessed by hematologic, renal, hepatic and coagulation parameters.

Exclusion Criteria:

1. Participant has a concomitant malignancy, or participant has a prior non-endometrial invasive malignancy who has been disease-free for <3 years or who received any active treatment in the last 3 years for that malignancy. Non-melanoma skin cancer is allowed.
2. Participant has any medical history of interstitial lung disease or pneumonitis.
3. Participant has cirrhosis or current unstable liver or biliary disease.
4. Participant has known uncontrolled central nervous system metastases, carcinomatosis meningitis, or both.
5. Participant has a diagnosis of immunodeficiency.
6. Participant has received prior therapy with an anti- Programmed death protein 1 (PD-1), anti- Programmed death ligand 1 (PD-L1), anti- Programmed death ligand 2 (PD-L2), or anti- Cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) agent.
7. Participant has not recovered adequately from AEs.
8. Participant has received prior anticancer therapy (chemotherapy, targeted therapies, hormonal therapy, radiotherapy, or immunotherapy) within 21 days prior to the first dose of study intervention.
9. Participant has received any live vaccine within 30 days of the first dose of study intervention. Vaccination against coronavirus disease 2019 (COVID-19) using vaccines that are authorized via the appropriate regulatory mechanisms are not exclusionary.
10. Participant has Hepatitis B surface antigen (HBsAg) positive, or Hepatitis C virus (HCV) Ribonucleic acid (RNA) positive at screening or within 3 months prior to the first dose of study intervention.
11. Participant is known human immunodeficiency virus (HIV) infection.
12. Participant is currently participating and receiving study intervention or has participated in a study of an investigational agent and received study intervention or used an investigational device within 4 weeks of the first dose of treatment.
13. Participant with contraindication to carboplatin and paclitaxel.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Durable Response Rate for 12 months (DRR12) assessed by Blinded Independent Central Review (BICR) | Up to approximately 148 weeks
  DRR12 is defined as the proportion of participants with confirmed Complete Response (CR) or Partial Response (PR), and Duration of Response (DOR) lasting greater than or equal to (≥) 12 months, per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
DRR12 assessed by Investigator | Up to approximately 148 weeks
  DRR12 is defined as the proportion of participants with confirmed Complete Response (CR) or Partial Response (PR), and Duration of Response (DOR) lasting greater than or equal to (≥) 12 months, per RECIST 1.1.
Progression-free survival (PFS) per RECIST 1.1, assessed by BICR | Up to 226 weeks
  PFS is defined as the time from the date of first dose to the date of first documented disease progression (PD) or death due to any cause, whichever comes first.
Progression-free survival (PFS) per RECIST 1.1, assessed by investigator | Up to 226 weeks
  PFS is defined as the time from the date of first dose to the date of first documented PD or death due to any cause, whichever comes first.
Overall survival (OS) | Up to 226 weeks
  OS is defined as time from first dose of study intervention to death from any cause.
Overall response rate (ORR) per RECIST 1.1 assessed by BICR | Up to 226 weeks
  ORR is defined as the proportion of participants with confirmed CR or PR.
ORR per RECIST 1.1 assessed by Investigator | Up to 226 weeks
  ORR is defined as the proportion of participants with confirmed CR or PR.
Duration of response (DOR) per RECIST 1.1 assessed by BICR | Up to 226 weeks
  DOR is defined as the time from the date of first documented objective response (confirmed CR or PR) to the date of first documented PD or death due to any cause, whichever comes first.
DOR per RECIST 1.1 assessed by Investigator | Up to 226 weeks
  DOR is defined as the time from the date of first documented objective response (confirmed CR or PR) to the date of first documented PD or death due to any cause, whichever comes first.
Serum concentration of dostarlimab | Up to 67 weeks
Concentration at the end of infusion (C-EOI) for dostarlimab | Up to 67 weeks
Trough concentration (Ctrough) for dostarlimab | Up to 67 weeks
Number of participants with Anti-drug antibody (ADA) against dostarlimab | Up to 226 weeks
Number of participants with adverse events (AEs), Immune-mediated adverse events (imAEs), and serious adverse events (SAEs) by severity | Up to 226 weeks
Number of participants with AEs, imAEs, and SAEs leading to dose modifications or study intervention discontinuation | Up to 226 weeks
Number of participants with AEs leading to death | Up to 226 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/